CLINICAL TRIAL: NCT03000699
Title: Efficacy of Cognitive Bias Modification in Residential Treatment for Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, Lena Quilty, Independent Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 077/2016
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Substance Dependence
Keywords: cognitive bias modification; interpretation bias; suicidal ideation; depression
MeSH Terms: conditions — Substance-Related Disorders; Suicidal Ideation; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Bias Modification (Experimental): 64 training paragraphs, approximately 10-20 seconds each, digitally recorded and presented stereophonically through headphones, delivered over the course of one week.
  Interventions: Behavioral: Cognitive Bias Modification
- Assessment-Only Control (No Intervention): No training will be provided.

INTERVENTIONS:
Behavioral: Cognitive Bias Modification — Training paragraphs describe scenarios designed to be ambiguous at the outset and to resolve in a positive direction, with the intention of establishing a learning contingency between the ambiguity at the beginning of the scenario and the positive resolution that becomes clear towards the end of the statement.
  Arms: Cognitive Bias Modification

SUMMARY:
The purpose of this study is to determine whether computer bias modification for interpretation bias (CBM-I) is effective in the reduction of suicidal ideation in substance use disorders.

DETAILED DESCRIPTION:
Eighty-eight adult inpatients completing residential treatment in the Addictions Services at the Centre for Addiction and Mental Health (CAMH) will be randomized to receive CBM-I daily for one week, adjunct to the residential psychosocial treatment or to an assessment-only control condition. Participants will complete clinical measures consisting of interviews and questionnaires measuring suicidal ideation, hopelessness, depression, negative affect, and interpretation biases before, during and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Exhibit moderate suicide risk or greater
* Be enrolled in the Addictions Services inpatient program
* Fluent in reading English
* Capacity to give informed consent

Exclusion Criteria:

* A lifetime diagnosis of a psychotic or bipolar disorder
* Significant neurological disorder or psychical illness likely to interfere with participation
* Psychotropic medication changes within the past two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Columbia-Suicide Severity Rating Scale, Screen Version (C-SSRS) | Seven days
  This scale quantifies the severity of suicidal ideation and behaviour.

SECONDARY OUTCOMES:
Beck Hopelessness Scale (BHS) | Seven days
  This questionnaire assesses thoughts and emotions associated with the future.
Beck Depression Inventory II (BDI-II) | Seven days
  This questionnaire assesses severity of depressive symptoms and cognitions.
Positive and Negative Affect Schedule (PANAS) | Seven days
  This questionnaire assesses current positive and negative mood
Scrambled Sentences Tests | Seven days
  This computer test will be used as an implicit measure of negative interpretation bias.

CONTACTS AND LOCATIONS:
Overall Officials: Lena C Quilty, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.ca/research